CLINICAL TRIAL: NCT01306435
Title: Effects of Low Power Laser Associated With Exercises in Osteoartite Knee: Randomized Clinical Trial, Double-blind, Controlled
Brief Title: Low Power Laser and Exercise in Osteoarthritis of the Knee: a Randomized Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Amélia Pasqual Marques, Departamnto Speech Therapy, Physiotherapy and Occupational Therapy, Faculty of Medicine, University of São Paulo, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 077508
Record Dates: First submitted 2011-02-23; First posted 2011-03-01 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Low Power Laser Therapy; Exercise; Knee
MeSH Terms: conditions — Osteoarthritis; Motor Activity | interventions — Lasers; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser Group (Experimental)
  Interventions: Other: Laser
- Placebo Group (Placebo Comparator)
  Interventions: Other: Placebo Laser

INTERVENTIONS:
Other: Laser — 3-week treatment with three Laser sessions per week
  Other Names: LOW POWER LASER
  Arms: Laser Group
Other: Placebo Laser — 3-week treatment with three Placebo Laser sessions per week
  Other Names: PLACEBO LOW POWER LASER
  Arms: Placebo Group

SUMMARY:
Indroduction: Knee osteoarthritis (OA) is a painful condition causing disability, weakness and poor quality of live. The results are very consistent about the benefits of laser and exercises to improve pain and function in subjects with knee osteoarthritis Objectives: To investigate the effects of Low Power Laser (LBP) associated with exercise in pain, function, range of motion, muscle strength and quality of life of patients with knee osteoarthritis.

Methods: Forty patients of both sexes aged between 50 and 75 years with knee osteoarthritis (grade 2-4) were randomized into two groups: Laser-LBP-active dose of 3J more exercises and Group Placebo-LBP- placebo and exercise. Were evaluated for pain, function, range of motion, muscle strength and quality of life on three occasions: before starting treatment (evaluation 1), 3 weeks after laser application (evaluation 2) and 8 weeks after completion of exercise (evaluation 3). There were 33 physical therapy sessions three times a week, on March 1 and the laser was applied in the other, only the exercises.

DETAILED DESCRIPTION:
Pain: Pain intensity was measured with the Visual Analogue Scale (VAS) which is a straight 10 cm long devoid of numbers, in which there is only an indication of the extreme left of "no pain" and extreme right to "unbearable pain". The higher the score, the greater the pain.

Feature: Survey conducted by Lequesne, which is an index composed of 11 questions about pain, discomfort and function. The scores range from 0 to 24 (without affecting the extremely severe, respectively), the higher the score, the greater the impairment.

Range of motion (ROM): ADM flexion and knee extension was measured using a universal goniometer (AESCULAP) with the patient prone second methodology Marques.

Muscular Strength: To assess the maximal isometric strength of the quadriceps muscle was used Dynamometer model Lafayette ® Portable (USA), while seated at 60 ° of knee flexion and this gradation was controlled with a goniometer. Patients remained seated on the stretcher and held steady with thigh extension strength, the dynamometer being maintained in the distal leg. Three measurements were taken, and the mean value.

Quality of Life: The Questionnaire was used Western Ontario and McMaster Universities Osteoarthritis (WOMAC)a self-assessment that evaluates pain, stiffness and physical activity. The higher the score, the greater the impact of OA on quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of osteoarthritis
* Knee pain
* Functional reduction in the last three months
* Grade 2-4 OA
* Fulfilled at least one of the classification criteria of the American College of Rheumatology

Exclusion Criteria:

* Cancer
* Diabetes mellitus
* Symptomatic hip OA
* Antidepressants
* Anti-inflammatory steroidal and nonsteroidal or tranquilizers in the last six months and throughout the treatment

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in VAS at 3 and 8 weeks | baseline, 3 and 8 weeks
  In the VAS the subject marks the intensity of its pain in a centimeter horizontal line

SECONDARY OUTCOMES:
Change from baseline in Lequesne at 3 an 8 weeks | baseline, 3 and 8 weeks
  Lequesne index is a composite of 11 questions about pain, discomfort and function. The scores range from 0 to 24 (without affecting the extremely severe, respectively), the higher the score, the greater the impairment.
Change from baseline in range of motion | baseline, 3 and 8 weeks
  ADM flexion and knee extension was measured using a universal goniometer (AESCULAP) with the patient prone
Change from baseline in Muscular Strength at 3 and 8 weeks | baseline, 3 and 8 weeks
  To assess the maximal isometric strength of the quadriceps muscle was used Dynamometer model Lafayette ® Portable (USA), while seated at 60 ° of knee flexion and this gradation was controlled with a goniometer. Patients remained seated on the stretcher and held steady with thigh extension strength, the dynamometer being maintained in the distal leg. Three measurements were taken, and the mean value
Change from baseline in Quality of Life at 3 and 8 weeks | baseline, 3 and 8 weeks
  The Questionnaire was used Western Ontario and McMaster Universities Osteoarthritis (WOMAC) a self-assessment that evaluates pain, stiffness and physical activity. The higher the score, the greater the impact of OA on quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Patrícia P Alfredo, MS, Principal Investigator — Faculty of Medicine of the University of São Paulo; Amélia P Marques, PhD, Study Director — Faculty of Medicine of the University of São Paulo
Locations (1):
- University of São Paulo General Hospital, São Paulo, São Paulo, Brazil